CLINICAL TRIAL: NCT04597918
Title: An Exploratory, Prospective, Multi-Center, Open-Label, Single-Arm, Interventional, Phase IIB Study to Investigate Aqueous Humor and Multimodal Imaging Biomarkers in Treatment-Naïve Patients With Diabetic Macular Edema Treated With Faricimab (RO6867461) - ALTIMETER STUDY
Brief Title: A Study to Investigate Aqueous Humor and Multimodal Imaging Biomarkers in Treatment-Naïve Participants With Diabetic Macular Edema Treated With Faricimab
Acronym: ALTIMETER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MR41926; 2020-001174-30 (EudraCT Number)
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Faricimab (Experimental): Participants will receive 6 doses (one 6 mg faricimab intravitreal [IVT] injection every 28 days [Q4W]) starting at Day 1 and ending on the Day 140 visit. Participants will return for a safety follow-up visit (SFV) after ≥28 days and within <35 days following their last study treatment.
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — A 6-milligram (mg) dose of faricimab will be administered intravitreally (IVT) in the study eye once every 4 weeks (Q4W).
  Other Names: VABYSMO™; RO6867461; RG7716

SUMMARY:
This is an exploratory, prospective, multicenter, open-label, single-arm, interventional, Phase IIb study designed to explore the associations over time between clinical assessments, multimodal imaging assessments, aqueous humor (AH) biomarker patterns, and genetic polymorphisms in participants with diabetic macular edema (DME) who are treated with faricimab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (Type 1 or Type 2), as defined by the World Health Organization (WHO) and/or American Diabetes Association
* Hemoglobin A1c (HbA1c) ≤10%
* Patients who are intravitreal (IVT) treatment-naïve in the study eye
* Diabetic macular edema (DME) defined as macular thickening by spectral-domain optical coherence tomography (SD-OCT) involving the center of the macula. This inclusion criterion is to be assessed by the central reading center (CRC).
* Decreased visual acuity (VA) attributable primarily to DME
* Clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images to confirm diagnosis

Exclusion Criteria:

* Currently untreated diabetes mellitus or previously untreated patients who initiated oral or injectable anti-diabetic medication within 3 months prior to Day 1
* Any known hypersensitivity to any of the components in the faricimab injection, dilating eye drops, or any of the anesthetics and antimicrobial preparations used by the patient during the study
* Any major illness or major surgical procedure within 1 month before the Day 1. One re-screening for this criterion is permitted
* History of other diseases, other non-diabetic metabolic dysfunction, physical examination finding, historical or current clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of the faricimab or that might affect interpretation of the results of the study or renders the patient at high-risk for treatment complications, in the opinion of the Investigator
* Active cancer within the past 12 months prior to Day 1 except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, and prostate cancer with a Gleason score of ≤6 and a stable prostate-specific antigen for >12 months
* Stroke or myocardial infarction within 12 months prior to the Day 1. One re-screening for this criterion is permitted
* Any febrile illness within 1 week prior to Day 1. One re-screening for this criterion is permitted
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of faricimab
* Renal failure requiring renal transplant, hemodialysis, or peritoneal dialysis within 6 months prior to Day 1 or anticipated to require hemodialysis or peritoneal dialysis at any time during the study
* Any condition resulting in a compromised immune system that is likely to impact the aqueous humor (AH) inflammatory biomarkers.
* Patients who are currently enrolled in or have participated in any other clinical study involving an investigational product or device, or in any other type of medical research, within 3 months or 5 half-lives prior to Day 1 and up to completion of the current study
* Substance abuse occurring within 12 months prior to screening, in the Investigator's judgment
* Use of systemic immunomodulatory treatments within 6 months or 5 half-lives prior to Day 1
* Use of any systemic corticosteroids (including inhaled corticosteroids from inhalers used regularly, e.g., pulmonary disease, asthma, or seasonal allergy) within 1 month prior to Day 1
* Any prior or concomitant systemic anti-VEGF treatment within 6 months or 5 half-lives prior to Day 1
* Use of systemic medications known to be toxic to the lens, retina or optic nerve used during the 6-month period or 5 half-lives prior to Day 1 or likely need to be used
* Received a blood transfusion within 3 months prior to the screening visit
* Received any treatment that leads to immunosuppression within 6 months or 5 half-lives prior to Day 1

Ocular Exclusion Criteria for Study Eye:

* High-risk PDR. This exclusion criterion is to be assessed by the CRC
* Any history of or ongoing rubeosis iridis
* Any panretinal photocoagulation or macular laser photocoagulation treatment received in the study eye prior to the screening visit or expected to be received between the screening visit and Day 1
* Any history of treatment with anti-VEGF or any periocular or IVT corticosteroids in the study eye and no such treatment planned for the time between screening and Day 1
* Any treatment for dry eye disease in the last month prior to Day 1. Lubricating eye drops and ointments are permitted.
* Any treatment with anti-inflammatory eye drops within 1 month prior to Day 1
* Any intraocular surgery within 3 months prior to Day 1 or any planned surgery during the study
* Any glaucoma surgery/laser procedure involving the iris, trabecular meshwork, or ciliary body prior to the screening visit. Only iris surgery/laser might be allowed if they occurred more than 6 months prior to Day 1.
* History of vitreoretinal surgery/pars plana vitrectomy, corneal transplant, or radiotherapy
* Any active or suspected ocular or periocular infections on Day 1
* Any presence of active intraocular inflammation on Day 1 or any history of intraocular inflammation
* Any history of idiopathic, infectious, or noninfectious uveitis
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision
* Any current ocular condition or other causes of visual impairment for which, in the opinion of the Investigator, VA loss would not improve from resolution of macular edema

Ocular Exclusion Criteria for Fellow Eye:

* Patient is currently receiving treatment with brolucizumab or bevacizumab in the non-study eye and is unwilling to switch to a protocol allowed non-study eye treatment during the study
* Any previous treatment with Iluvien® or Retisert® in the non-study eye
* Non-functioning non-study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (12):
  - Bascom Palmer Eye Institute, Naples, Florida
  - Northwestern Medical Group/Northwestern University, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - The Retina Institute, St Louis, Missouri
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
- Argentina (2):
  - Centro Oftalmológico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
- Canada (2):
  - Vitreous Retina Macula Specialists of Toronto, Etobicoke, Ontario
  - The Retina Centre of Ottawa, Ottawa, Ontario
- Universitätsklinikum Tübingen, Tübingen, Germany
- Italy (2):
  - Ospedale San Giuseppe; U.O. Oculistica, Milan, Lombardy
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
- Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Warsaw, Poland
- United Kingdom (3):
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Kings College Hospital, London
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 99 patients were enrolled in the study at 23 sites in 7 countries.
Groups:
- Faricimab: Participants received 6 doses of faricimab (one 6-mg faricimab intravitreal [IVT] injection every 28 days [Q4W]) starting at Day 1 and ending on the Day 140 visit. Participants returned for a safety follow-up visit (SFV) after ≥28 days and within <35 days following their last study treatment.
Period: Overall Study
Arm/Group | Faricimab
Started | 99
Completed | 89
Not Completed | 10
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: There were 2 analysis populations in this study, the modified intent-to-treat (mITT; all patients enrolled in the study that received any amount of study treatment) and safety-evaluable (SAF; all patients enrolled in the study who received at least 1 injection of study treatment) populations. All 99 participants were included in both the mITT and SAF populations.
Arm/Group | Faricimab
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 7
  White | 86
  Asian | 5
  Unknown | 1
Region of Enrollment [Count of Participants; unit: Participants]
  US and Canada | 62
  Rest of the World | 37
Best-Corrected Visual Acuity (BCVA) in the Study Eye at Baseline [Mean (Standard Deviation); unit: ETDRS Letters] — Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score).
  ETDRS Letters | 62.5 (11.8)
Central Subfield Thickness (CST) in the Study Eye at Baseline [Mean (Standard Deviation); unit: microns] — Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using Spectral Domain-Optical Coherence Tomography (SD-OCT).
  microns | 464.0 (149.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥2-Step Improvement From Baseline on the Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS) in the Study Eye at Week 24
Description: The ETDRS DRSS score of each participant's study eye was assessed using ultra-wide field color fundus photography (UWF-CFP) taken by trained personnel at the study sites. Analysis of the fundus photographs was performed by the central reading center, and the percentage of participants with a ≥2-step improvement from baseline was summarized along with a two-sided 95% Clopper-Pearson exact confidence interval. Baseline was defined as the participant's last observation prior to initiation of study drug.
Time Frame: Baseline and Week 24
Population: Participants in the modified intent-to-treat (mITT) Population with missing baseline assessments were excluded from the analysis. The number analyzed indicates participants with assessments at both Baseline and Week 24.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Faricimab
Number analyzed (Participants) | 64
Percentage of participants | 50.0 [37.2 to 62.8]

2. Secondary Outcome: Adjusted Mean Change From Baseline in Best-Corrected Visual Acuity (BCVA) in the Study Eye at Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. For the Mixed Model for Repeated Measures (MMRM) analysis, the model adjusted for visit, age (continuous), baseline BCVA (continuous), and region (US and Canada and the rest of the world). An unstructured covariance structure was used. In case of convergence issues with the model, an AR (1) covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM.
Time Frame: From Baseline to Week 24
Population: The modified intent-to-treat (mITT) population is defined as all participants enrolled in the study that received any amount of study treatment.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Faricimab
Number analyzed (Participants) | 99
ETDRS Letters | 9.2 [7.5 to 10.9]

3. Secondary Outcome: Adjusted Mean Change From Baseline in Central Subfield Thickness in the Study Eye at Week 24
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using Spectral Domain-Optical Coherence Tomography (SD-OCT), as assessed by the central reading center. For the Mixed Model of Repeated Measures (MMRM) analysis, the model was adjusted for visit, age (continuous), baseline CST (continuous), and region (US and Canada and the rest of the world). An unstructured covariance structure was used. In case of convergence issues with the model, an AR (1) covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM.
Time Frame: From Baseline to Week 24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Faricimab
Number analyzed (Participants) | 99
microns | -200.2 [-214.1 to -186.2]

4. Secondary Outcome: Median Time to First Absence of DME in the Study Eye During the Study
Description: An event was defined as the first absence of diabetic macular edema (DME) in the study eye, defined as first time reaching central subfield thickness (CST; ILM-RPE) <305 microns, after baseline. Baseline was defined as the participant's last observation prior to initiation of study drug. The time to first absence of DME was a Kaplan-Meier estimate. The 95% confidence interval (CI) for the median was computed using the method of Brookmeyer and Crowley. Participants without an event and discontinued from treatment were censored at the last CST assessment.
Time Frame: From Baseline to Week 24
Population: The modified intent-to-treat (mITT) population is defined as all participants enrolled in the study that received any amount of study treatment. Participants with absence of DME at Baseline were excluded from the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Faricimab
Number analyzed (Participants) | 98
Weeks | 8.0 [8.0 to 12.0]

5. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye at Week 24
Description: The absence of intraretinal fluid (IRF) in the study eye (defined as IRF absent or definite outside center subfield only) was assessed by the central reading center using Spectral Domain-Optical Coherence Tomography (SD-OCT). The percentage of participants with absence of IRF and a two-sided 95% Clopper-Pearson exact confidence interval are reported.
Time Frame: Week 24
Population: Participants in the modified intent-to-treat (mITT) Population with non-missing Week 24 assessments were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Faricimab
Number analyzed (Participants) | 88
Percentage of participants | 26.1 [17.3 to 36.6]

6. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye at Week 24
Description: The absence of subretinal fluid (SRF) in the study eye (defined as SRF absent or definite outside center subfield only) was assessed by the central reading center using Spectral Domain-Optical Coherence Tomography (SD-OCT). The percentage of participants with absence of SRF and a two-sided 95% Clopper-Pearson exact confidence interval are reported.
Time Frame: Week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Faricimab
Number analyzed (Participants) | 88
Percentage of participants | 98.9 [93.8 to 100.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until ≥28 days to <35 days after the last dose of study drug (up to 24 weeks)
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received at least one injection of faricimab in the study eye. For ocular AEs, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Arm/Group | Faricimab
All-Cause Mortality (participants affected / at risk) | 1/99
Serious Adverse Events (participants affected / at risk) | 8/99
Other Adverse Events (participants affected / at risk) | 21/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faricimab (N=99)
Localised infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Spinal operation (Surgical and medical procedures) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faricimab (N=99)
Diabetic retinal oedema (Eye disorders) | 6 (6)
Retinal exudates (Eye disorders) | 5 (10)
COVID-19 (Infections and infestations) | 7 (7)
Hypertension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04597918/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT04597918/SAP_001.pdf